CLINICAL TRIAL: NCT03227432
Title: An Exploratory Study to Evaluate the Combination of Elotuzumab and Nivolumab With and Without Pomalidomide in Relapsed Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn before enrollment due to issues around the FDA hold on PD-1/PD-L1 drugs in combination with IMIDs.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jacob Laubach, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-645
Record Dates: First submitted 2017-07-07; First posted 2017-07-24 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; pomalidomide; elotuzumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab + Elotuzumab (Experimental): * 22 patients will be entered, If > 4 patients achieve at least a partial response (PR) within 4 cycles an additional 18 patients will be treated.
  * Nivolumab will be administered intravenously twice per cycle for cycle 1-4
  * Nivolumab will be administered intravenously once per cycle for cycle 5
  * Elotuzumab will be administered intravenously 4 times per cycle for cycle 1-2
  * Elotuzumab will be administered intravenously twice per cycle for cycle 3-4
  * Elotuzumab will be administered intravenously once per cycle for cycle 5
  Interventions: Drug: Elotuzumab; Drug: Nivolumab
- Nivolumab+Elotuzumab+Pomalidomide+Dexamethasone (Experimental): * Nivolumab will be administered intravenously twice per cycle for cycle 1-4
  * Nivolumab will be administered intravenously once per cycle for cycle 5
  * Elotuzumab will be administered intravenously 4 times per cycle for cycle 1-2
  * Elotuzumab will be administered intravenously twice per cycle for cycle 3-4
  * Elotuzumab will be administered intravenously once per cycle for cycle 5
  * Pomalidomide will be administered for 21 days per cycle
  * Dexamethasone will be administered weekly
  Interventions: Drug: Dexamethasone; Drug: Pomalidomide; Drug: Elotuzumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone, a corticosteroid, is similar to a natural hormone produced by adrenal glands. It relieves inflammation.
  Other Names: Maxidex
  Arms: Nivolumab+Elotuzumab+Pomalidomide+Dexamethasone
Drug: Pomalidomide — Pomalidomide which is an immunomodulatory drug. This means that pomalidomide modulates the immune system to help fight diseases.
  Other Names: Pomalyst
  Arms: Nivolumab+Elotuzumab+Pomalidomide+Dexamethasone
Drug: Elotuzumab — Elotuzumab is an antibody, that stimulates the immune system to fight diseases
  Other Names: Empliciti
Drug: Nivolumab — Nivolumab works by blocking an inhibitory signal within immune cells, potentially allowing the immune system to fight the cancer
  Other Names: Opdivo

SUMMARY:
This research study is studying a combination of targeted therapies as a possible treatment for multiple myeloma (MM).

The drugs involved in this study are:

* Elotuzumab
* Nivolumab
* Pomalidomide
* Dexamethasone

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug combination to learn whether the combination works in treating a specific disease. "Investigational" means that the drug combination is being studied.

This study has two parts. Each part tests a different combination of drugs.

* In Part 1 participants will be given elotuzumab and nivolumab.
* In Part 2 participants will be given elotuzumab, nivolumab, pomalidomide, and dexamethasone.

Each of these drugs works in a different way to help the body fight multiple myeloma. The drugs are being tested in different combinations to see if they are more effective when taken together.

Elotuzumab is an antibody, that stimulates the immune system to fight your disease. The FDA (the U.S. Food and Drug Administration) has approved elotuzumab in combination with lenalidomide as a treatment option for this disease.

In this research study, the participant will receive pomalidomide which is an immunomodulatory drug. This means that pomalidomide modulates the immune system to help fight the disease. The FDA has approved pomalidomide as a treatment option for this disease after receiving two other therapies.

Dexamethasone, also FDA approved, is a type of steroid and is usually combined with other chemotherapy for the treatment of blood cancers, such as myeloma and leukemias.

The FDA has not approved nivolumab for this specific disease but it has been approved for other uses, specifically lung cancer. Nivolumab works by blocking an inhibitory signal within immune cells, potentially allowing the immune system to fight the cancer.

In this research study the investigators are looking to see if the combination of elotuzumab, nivolumab, pomalidomide, and dexamethasone is effective in fighting the cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥ age 18 years
* Patient is able to understand and has given voluntary written informed consent before performance of any study-related procedures not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care
* Patient has been previously diagnosed with MM based on standard International Myeloma Working Group (IMWG) criteria and currently requires treatment.
* Patient must have received at least two previous lines of therapy for multiple myeloma including lenalidomide or thalidomide and a proteasome inhibitor (bortezomib, carfilzomib or ixazomib).
* Patient must have demonstrated disease progression on or within 60 days of completion of the last therapy. Patient has measurable disease defined as at least one of the following:

  * Serum M protein ≥ 0.5 g/dL (≥5 g/L)
  * Urine M protein ≥200 mg/24 hours
  * Serum free light chain (FLC) assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Appendix A)
* Negative serum or urine pregnancy test for women of child-bearing potential
* Screening Laboratory parameters:
* Absolute neutrophil count (ANC) ≥ 1,000 cells/dL (1.0 x 109/L). Granulocyte colony-stimulating factor (GCSF) is not permitted during screening to meet eligibility criteria and within 14 days of initiation of therapy

  * Platelet count ≥ 75,000 cells/dL (75 x 109/L) Platelet transfusion is not permitted during screening to meet eligibility criteria and within 14 days of initiation of therapy
  * Hemoglobin ≥ 8.0 g/dl ( red blood cell (RBC) transfusions are permitted during the screening period)
  * Total Bilirubin ≤ 1.5 X upper limit of normal (ULN) (Patients with known Gilbert Syndrome are allowed to have total bilirubin < 3.0 mg/dL)
  * Aspartate transaminase (AST, or SGOT) and alanine transaminase (ALT, or SGPT) ≤ 3.0x ULN
  * Estimated creatinine clearance by Cockcroft-Gault formula ≥ 40 mL/min
  * Serum creatinine < 1.5 X ULN. (Appendix C)

Exclusion Criteria:

* Diagnosed or treated for another malignancy within 3 years prior to enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low risk prostate cancer after curative therapy.
* Prior therapy with pomalidomide
* Prior treatment with monoclonal antibodies including elotuzumab
* Prior therapy with anti-programmed death 1 (PD-1) or programmed death-ligand 1 (PD-L1) agents.
* Received any investigational drug within 14 days or 5 half-lives of the investigational drug, whichever is longer.
* Prior anti-cancer therapy within 14 days.
* Patient has any Grade 3 or > unresolved adverse reaction from previous treatment. Previous allogeneic stem cell transplantation with active graft-versus-host disease (GVHD) or being under immunosuppressive therapy in the last 2 months prior to inclusion in the trial.
* Autologous stem cell transplant if < 12 weeks from enrollment.
* Daily requirement for oral corticosteroids (equivalent to > 10 mg/day prednisone daily) Inhaled or topical corticosteroids are allowed.
* Patient is human immunodeficiency virus (HIV) positive,.
* Patient is Hepatitis B Surface antigen-positive.
* Patient has active hepatitis C infection.
* Patient has an autoimmune disease. (Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger).
* Any clinically significant, uncontrolled medical conditions that, in the treating Investigator's opinion, would impose excessive risk to the patient or may interfere with compliance or interpretation of the study results. Uncontrolled intercurrent illness may include, but is not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations as determined by treating investigator that would limit compliance with study requirements.
* History of erythema multiforme or severe hypersensitivity to prior IMiD's®
* Inability to tolerate thromboprophylaxis
* Known severe intolerance to prior steroid therapy (Grade 3 or above adverse event which was unresponsive to a dose reduction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response Rate | 2 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 months

SECONDARY OUTCOMES:
The Rate of Clinical Benefit Response (CBR) | 2 years
Time to Response | 2 years
Duration of Response | 2 years
Progression Free Survival | 2 years
Overall Survival | 2 years
Time to Treatment Failure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Laubach, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No